CLINICAL TRIAL: NCT02650557
Title: Prediction Value of Ecg on Coronary Slow-flow (PECS) Study
Brief Title: Prediction Value of Ecg on Coronary Slow-flow
Acronym: PECS
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, department of cardiology, first affiliated hoapital of SYSU, Sun Yat-sen University
Other Study IDs: PECS-sysu
Record Dates: First submitted 2016-01-03; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Slow Flow
Keywords: coronary slow flow; P-wave dispersion
MeSH Terms: interventions — Cerebral Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CSF group: consecutive patients with angiographically documented CSF
  Interventions: Procedure: angiography
- control group: age- and gender-matched control subjects
  Interventions: Procedure: angiography

INTERVENTIONS:
Procedure: angiography — angiography or arteriography is a medical imaging technique used to visualize the inside, or lumen, of blood vessels and organs of the body, with particular interest in the arteries, veins, and the heart chambers. This is traditionally done by injecting a radio-opaque contrast agent into the blood vessel and imaging using X-ray based techniques such as fluoroscopy.

SUMMARY:
The investigators aimed to investigate the vessel heterogeneity of Thrombolysis in Myocardial Infarction frame count (TFC) in the three coronary arteries, and its relation to P-wave dispersion, in patients with coronary slow flow and otherwise normal coronary arteries.

DETAILED DESCRIPTION:
Coronary slow flow (CSF) phenomenon, which is characterized by delayed coronary opacification in the absence of obstructive epicardial coronary artery disease, is a relatively common finding in patients undergoing routine coronary angiography and is often associated with chest pain. In some patients with CSF, blood flow may be heterogeneously distributed in the three coronary arteries, suggesting the heterogeneously distributed microvascular dysfunction in the myocardium. However, the vessel heterogeneity of Thrombolysis in Myocardial Infarction (TIMI) frame count (TFC) has not been fully elucidated.

P-wave dispersion (PWD) is defined as the difference between the longest and the shortest P-wave duration recorded from multiple different surface electrocardiogram (ECG) leads, and it has been reported to be associated with inhomogeneous and discontinuous propagation of sinus impulses5, which are well known electrophysiologic characteristics of the atrium prone to fibrillation. Although it is plausible to hypothesize that PWD might be associated with the heterogeneously distributed microvascular dysfunction, and previous studies have demonstrated the abnormal PWD in patients with CSF, the correlation between TFC heterogeneity and PWD has never been evaluated.

In this study, the investigators aimed to investigate the vessel heterogeneity of TFC in the three coronary arteries, and its relation to PWD, in patients with CSF and otherwise normal coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* All of the subjects had chest pain and were referred to our catheterization laboratory for coronary angiography

Exclusion Criteria:

* Valvular or congenital heart disease
* Atrial fibrillation or other arrhythmia that would interfere with ECG analysis
* Left ventricular hypertrophy
* Myocardial or pericardial disease
* Chronic obstructive pulmonary disease, or electrolyte abnormalities.
* Subjects taking antiarrhythmic, antiischemic, β-blocker, or calcium-channel blocker medications were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the subjects had chest pain and were referred to our catheterization laboratory for coronary angiography. Diagnosis of CSF was based on thrombolysis in myocardial infarction (TIMI) frame count (TFC).
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Average thrombolysis in myocardial infarction (TIMI) frame count (TFC) in the three coronary arteries and its relation to P waves parameters on ECG in patients with CSF and otherwise normal coronary arteries | 24-72 hours
  The first frame was defined as the frame in which concentrated dye occupies the full width of the proximal coronary artery lumen, touching both borders of the lumen, and indicates forward motion down the artery. The final frame counted is that in which the contrast first reaches the distal predefined landmark branch without the necessity for full opacification. The difference between maximum and minimum P wave duration (Pmax and Pmin) was calculated from the 12-lead ECG and defined as PWD.

SECONDARY OUTCOMES:
maximum and minimum P wave duration (Pmax and Pmin) and major adverse cardiac events (MACE) in patients with CSF and otherwise normal coronary arteries | 24 hours-30 days
  The occurrence of major adverse cardiac events, defined as (1) death, (2) nonfatal myocardial infarction, or (3) target vessel revascularization. Myocardial infarction was diagnosed by a rise in the creatine kinase level to more than twice the upper normal limit with an increased creatine kinase-MB. Target lesion revascularization was defined as a repeat intervention (surgical or percutaneous) to treat a luminal stenosis within the stent or in the 5-mm distal or proximal segments adjacent to the stent. Target vessel revascularization was defined as a reintervention driven by any lesion located in the same epicardial vessel. Thrombotic stent occlusion was angiographically documented as a complete occlusion (TIMI flow 0 or 1) or a flow-limiting thrombus (TIMI flow 1 or 2) of a previously successfully treated artery.

CONTACTS AND LOCATIONS:
Overall Officials: zhimin du, MD, Principal Investigator — fitst affiliated hospital of SYSU
Locations (1):
- Xiaodong Zhaung, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No